CLINICAL TRIAL: NCT01056055
Title: Outcomes of the Modified-Brostrom Procedure Using Suture Anchor for Chronic Lateral Ankle Instability - A Prospective, Randomized Comparison With the Bone Tunnel Technique
Brief Title: Outcomes of the Modified-Brostrom Procedure Using Suture Anchor for Chronic Lateral Ankle Instability
Status: Completed | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Byung-Ki Cho, Chungbuk National University Hospital
Other Study IDs: titanick25; ClinicalTrials (Registry Identifier: ClinicalTrials)
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2007-03

CONDITIONS: Chronic Ankle Instability
Keywords: Ankle; Chronic lateral instability; Modified Brostrom procedure; Suture anchor; Bone tunnel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suture anchor, Bone tunnel: Suture anchor group: patients who underwent the modified Brostrom procedure using suture anchor technique Bone tunnel group: patients who underwent the modified Brostrom procedure using bone tunnel technique

SUMMARY:
This prospective, randomized study was conducted to compare the clinical outcomes of the modified Brostrom procedure using a suture anchor and bone tunnel for chronic lateral ankle instability.

DETAILED DESCRIPTION:
With With the increased number of participants in sports and leisure time activities, the incidence of ankle ligament injuries has been correspondingly increased. Various surgical methods have been reported for chronic ankle instability. Of these methods, the modified Brostrom procedure is currently used most frequently, and its excellent treatment outcomes have been reported. If there are any methods for obtaining a strong ligament fixation force which are both technically simple and safe, such methods would shorten the operative time and be helpful for surgeons with little experience in managing chronic ankle instability to obtain excellent treatment outcomes. In recent years, a procedure using a suture anchor, which is used for various types of ligament or tendon reconstructions, has been frequently performed. To date, however, few studies have reported clinical outcomes of suture anchor techniques and comparisons of clinical results between suture anchor techniques and other procedures. Given the above background, we prospectively compared the clinical outcomes between the bone tunnel and suture anchor techniques in the modified Brostrom procedure for chronic lateral ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complained of subjective instability of the ankle joint in whom repeated sprain injuries for > 6 months and pain were confirmed
* Patients with marked ankle instability confirmed by the anterior drawer test as compared with the contralateral ankle joint and tenderness involving the lateral ligament of the ankle joint was confirmed on physical examination
* Patients with an talar tilt angle exceeding 10o or a discrepancy of > 5o as compared with the non-affected side on stress radiography
* Patients with an anterior talar translation exceeding 10 mm or a discrepancy > 3 mm as compared with the non-affected side.

Exclusion Criteria:

* Patients who concurrently had an ankle fracture or marked tendon damage were excluded from the current analysis.

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Of patients who underwent the modified Brostrom procedure under the diagnosis of chronic lateral ankle instability, 40 patients (40 ankles) who could be followed during a minimum period of 2 years were enrolled in the current study. The current study included patients who complained of unilateral ankle joint instability.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The clinical evaluation consisted of a VAS for pain, the Karlsson scale, and the Sefton grading system. | during a minimum period of 2 years

SECONDARY OUTCOMES:
Talar tilt and anterior talar translation were measured on anterior and varus stress radiographs. | during a minimum period of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Ki Cho, M.D., Study Chair — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea